CLINICAL TRIAL: NCT06662097
Title: Multicenter Open-Label Feasibility Study of Intraoperative Nerve and Ureter Visualization With Bevonescein in Patients Undergoing Minimally Invasive Abdominopelvic Surgery
Brief Title: A Study of Bevonescein in Patients Undergoing Abdominopelvic Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alume Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ALM-488-004
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Surgery; Nerve Injury; Imaging

STUDY DESIGN:
Intervention Model Description: The study will begin with a dose-defining stage in each surgical setting. Once dose defining is complete, the study will proceed to a dose expansion phase for each surgical setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Defining (Experimental): A dose defining phase for each surgical setting.
  Interventions: Drug: Bevonescein
- Dose Expansion (Experimental): A dose expansion phase for each surgical setting.
  Interventions: Drug: Bevonescein

INTERVENTIONS:
Drug: Bevonescein — Bevonescein is a sterile solution that is intravenously administered
  Other Names: ALM-488

SUMMARY:
Feasibility study of Bevonescein to highlight Nerves and Ureter in patients undergoing Minimally Invasive Surgery

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability and efficacy of Bevonescein administered as an intravenous (IV) infusion to patients undergoing minimally invasive surgery. This study will also characterize the pharmacokinetic of Bevonescein in this subject population and determine the dose of Bevonescein needed to generate a fluorescence signal in nerve and ureter tissue to enable fluorescence recordings and image analysis with an imaging system.

ELIGIBILITY:
Inclusion Criteria:

* Must be a minimum of 18 years of age
* Study participant is planning to proceed with surgery
* Willing to provide informed consent
* Sexually active patients must be willing to use an acceptable form of contraceptive while participating and 30 days after.
* Females of childbearing potential must have a negative pregnancy test at screening and during the study.

Exclusion Criteria:

* Patient has had prior surgery at the intended surgical site.
* Patient has abnormal cardiac rhythm not controlled by medication.
* Patient has moderate to severe renal impairment.
* Patient has a history of fluorescein allergy.
* Patient has a history of drug-related anaphylactic.
* Presence of a concurrent disease or condition that may interfere with study participation.
* Presence or history of any condition that, in the view of the investigator, places the patient at high risk of treatment compliance.
* Use of any Investigational Product or investigational medial device within 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Fluorescence System Survey | 28 (+5 days)
  To assess the feasibility of the Fluorescence System in each of the identified Minimally Invasive Surgery settings.

SECONDARY OUTCOMES:
To determine the optimal dose of Bevonescein in Minimally Invasive Surgery settings | 28 (+5 days)
  The optimal dose for each of the identified surgical settings will be assessed by using three doses.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No